CLINICAL TRIAL: NCT00038792
Title: A Phase I/II Trial of Recombinant Human Keratinocyte Growth Factor (rHuKFG) for the Treatment of Steroid Refractory Gastrointestinal Acute Graft-versus-host Disease (aGvHD)
Brief Title: Phase I/II Trial rHuKFG for the Treatment of Steroid Refractory Gastrointestinal Acute GVHD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-036
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Acute Graft Versus Host Disease; Refractory
MeSH Terms: interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aGvHD (Experimental)
  Interventions: Drug: Recombinant Human Keratinocyte Growth Factor

INTERVENTIONS:
Drug: Recombinant Human Keratinocyte Growth Factor

SUMMARY:
Phase II efficacy evaluation, phase I/II efficacy and toxicity trial of recombinant human keratinocyte growth factor for the treatment of steroid refractory gastrointestinal graft versus host disease.

DETAILED DESCRIPTION:
There are two processes that cause diarrhea as the clinical manifestation of graft versus host disease. The first is the obvious immunologic attack on the colonic epithelium of the recipient. Once this immunologic attack has been abated the recipient is left with a colonic mucosa that is devoid of microvilli and has a smooth intestinal boarder. This is frequently subject to superinfections from bacteria all of which cause the diarrhea to continue. Researchers only endpoint to measure clinical response of immunosuppression is the resolution of diarrhea. The human recombinant keratinocyte growth factor stimulates the growth of colonic epithelium. The growth of colonic epithelium will in turn probably ameliorate some of the diarrhea associated with graft versus host disease.

ELIGIBILITY:
Inclusion criteria:

* Patients post allogeneic bone marrow transplant with watery diarrhea progressed on 2mg/kg of steroids after 3 days or failed to improve after 5 days.
* Patients may have skin or liver involvement with graft versus host disease.
* Patients should not have any infections etiology for diarrhea.

Exclusion criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2000-10; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with resolution of diarrhea | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James L. Gajewski, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org